CLINICAL TRIAL: NCT01808989
Title: Multicentric Study of the Clinical Interest of the TcPO2 Technique
Brief Title: Clinical Interest of the TcPO2 Technique
Acronym: CINEYSOFT
Status: Terminated | Type: Observational
Why Stopped: end of inclusing period
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2013-A00013-42
Record Dates: First submitted 2013-03-07; First posted 2013-03-12 (Estimated); Last update posted 2022-10-24 (Actual); Status verified 2022-10

CONDITIONS: Claudication
Keywords: peripheral artery disease; tcpo2; treadmill walking test; intermittent claudication
MeSH Terms: conditions — Intermittent Claudication; Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Exercise oxymetry

SUMMARY:
The measurement of the transcutaneous oxygen pressure records simultaneously the tcpO2 at the buttocks and chest level during walking. Before and after exercise the diagnosis, investigations and treatments ongoing or to be performed are recorded.

The present study focuses on the clinical interest of the transcutaneous oxygen pressure during exercise in the diagnosis of claudication in patient referred for an oximetry exercise test.

DETAILED DESCRIPTION:
Pre-test diagnostic hypothesis with probability will be completed by the physician.

Pre-test and post test ongoing or scheduled treatments will be completed by the physician.After the test, the same post test items will be evaluated.

Analysis will be done on differences of pre and post test results.

ELIGIBILITY:
Inclusion Criteria:

* referred for an oximetry exercise test
* Patient able to walk on a treadmill
* Patient covered by the French health insurance
* Patient able to understand the protocol
* Patient agrees to be involve in the protocol and sign the consent form

Exclusion Criteria:

* any heart issues during the last 3 months
* pregnancy

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with buttock pain and referred for an oximetry exercise test
Sampling Method: Non-Probability Sample
Enrollment: 952 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2022-10 (Actual); Study Completion 2022-10 (Actual)

PRIMARY OUTCOMES:
The percentage of patients for whom results tcpO2 effort led to changes in diagnosis measured by the questionnaire filled by the doctor in charge of the patient before and after the test | up to 1 day
  during a walk on a treadmill, there is a DROP of tcpo2<-15

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Abraham, MD; PhD, Principal Investigator — University hospital, Angers, FRANCE
Locations (8):
- France (8):
  - University Hospital, Angers
  - University Hospital, Lille
  - University Hospital, Lomme
  - University Hospital, Marseille
  - University Hospital, Nantes
  - University Hospital, Rennes
  - University Hospital, Toulouse
  - Hospital, Tours